CLINICAL TRIAL: NCT05850689
Title: A Randomized, Double-Blind, Placebo-controlled Multicenter Study to Assess the Efficacy and Safety of Lumateperone as Adjunctive Therapy in the Treatment of Patients With Major Depressive Disorder
Brief Title: Study of Lumateperone as Adjunctive Therapy in the Treatment of Patients With Major Depressive Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ITI-007-505
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder
Keywords: Adjunctive MDD Therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lumateperone 42 mg (Experimental)
  Interventions: Drug: Lumateperone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lumateperone — Lumateperone 42 mg capsules administered orally, once daily
  Arms: Lumateperone 42 mg
Drug: Placebo — Matching capsules administered orally, once daily
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled parallel-group, fixed-dose study in patients with a primary diagnosis of MDD according to criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) who have an inadequate response to ongoing ADT.

DETAILED DESCRIPTION:
The study will be conducted in three periods:

* Screening Period (up to 2 weeks) during which patient eligibility will be assessed.
* Double-blind Treatment Period (6 weeks) in which all patients will be randomized to receive placebo or lumateperone 42 mg/day in 1:1 ratio.
* Safety Follow-up Period (1 week) in which all patients will return to the clinic for a safety follow-up visit approximately one week after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the ages of 18 and 65 years, inclusive;
2. Meets DSM-5 criteria for MDD (MDD with psychotic features will be acceptable) as confirmed by the Investigator or Sponsor-approved rater using the modified Structured Clinical Interview for DSM-5, Clinical Trials Version (SCID-5-CT) and meets all of the following criteria:

   1. The start of the current major depressive episode (MDE) is at least 12 weeks but not more than 18 months prior to Screening;
   2. Has at least moderate severity of illness based on rater-administered MADRS total score ≥ 24 at Screening and at Baseline;
   3. Has at least moderate severity of illness based on CGI-S score ≥ 4 at Screening and at Baseline;
   4. Has a Quick Inventory of Depressive Symptomatology-Self Report-16 item (QIDS-SR-16) score ≥ 14 at Screening and at Baseline;
   5. Has sufficient history and medical record confirmation verifying the ADT and the current MDE is causing clinically significant distress or impairment in social, occupational, or other important areas of functioning.
3. Currently having an inadequate response (less than 50% improvement) to 2 or more ADTs in the current MDE as confirmed by the Investigator using the Antidepressant Treatment Response Questionnaire (ATRQ) and taking at least the minimum effective dose (per package insert) of one of the following antidepressants as monotherapy treatment for at least 6 weeks duration:

   1. citalopram/escitalopram
   2. fluoxetine
   3. paroxetine
   4. sertraline
   5. duloxetine
   6. levomilnacipran/milnacipran (if locally approved for MDD)
   7. venlafaxine/desvenlafaxine
   8. bupropion
   9. vilazodone
   10. vortioxetine

Exclusion Criteria:

1. Within the patient's lifetime, has a confirmed DSM-5 psychiatric diagnosis other than MDD, including:

   1. Schizophrenia, Schizoaffective Disorder, Schizophreniform Disorder or other psychotic disorder;
   2. Bipolar Disorder;
2. Within 6 months of Screening, has a confirmed DSM-5 psychiatric diagnosis other than MDD including:

   1. Anxiety disorders such as Panic Disorder or Generalized Anxiety Disorder; Obsessive-compulsive Disorder; Posttraumatic Stress Disorder as primary diagnoses. Note: Anxiety symptoms may be allowed if secondary to MDD, provided these symptoms do not require concurrent treatment;
   2. Eating disorder;
   3. Substance use disorders (excluding nicotine);
   4. Personality disorder of sufficient severity to have a major impact on the patient's psychiatric status;
   5. Within 12 months of Screening, has had any other psychiatric condition (other than MDD) that has been the main focus of treatment;
3. The patient experiences a ≥ 25% decrease in the MADRS total score between Screening and Baseline;
4. The patient experiences a ≥ 25% decrease in the QIDS-SR-16 total score between Screening and Baseline;
5. In the opinion of the Investigator, the patient has a significant risk for suicidal behavior during participation in the study or:

   1. At Screening, the patient scores "yes" on Suicidal Ideation Items 4 or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) within 6 months prior to Screening, or at Baseline, the patient scores "yes" on Suicidal Ideation Items 4 or 5 since the Screening Visit;
   2. At Screening, the patient has had 1 or more suicide attempts within 2 years prior to Screening;
   3. At Screening or Baseline, the patient scores ≥ 5 on MADRS Item 10 (Suicidal Thoughts), or
   4. The patient is considered to be in imminent danger to him/herself or others.
6. The patient has a first MDE at age 60 years or older.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | Day 43
  The MADRS is a clinician-rated 10 item scale to assess depressive symptoms. Each item is rated on a 7-point scale from 0-6. The total score ranges from 0 to 60 with a higher score indicating increased severity of depressive symptoms.

SECONDARY OUTCOMES:
Clinical Global Impression Scale-Severity | Day 43
  The CGI-S is a clinician-rated scale to assess a patient's overall mental health. The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).

CONTACTS AND LOCATIONS:
Locations (53):
- United States (21):
  - Clinical Site, Huntsville, Alabama
  - Clinical Site, Pico Rivera, California
  - Clinical Site, Farmington, Connecticut
  - Clinical Site, Clermont, Florida
  - Clinical Site, Hialeah, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Tampa, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Decatur, Georgia
  - Clinical Site, Kansas City, Kansas
  - Clinical Site, Overland Park, Kansas
  - Clinical Site, Methuen, Massachusetts
  - Clinical Site, O'Fallon, Missouri
  - Clinical Site, New York, New York
  - Clinical Site, Avon Lake, Ohio
  - Clinical Site, Cincinnati, Ohio
  - Clinical Site, Columbus, Ohio
  - Clinical Site, Philadelphia, Pennsylvania
  - Clinical Site, Houston, Texas
  - Clinical Site, Richardson, Texas
  - Clinical Site, Bellevue, Washington
- Bulgaria (6):
  - Clinical Site, Cherven Bryag
  - Clinical Site, Kardzhali
  - Clinical Site, Pleven
  - Clinical Site, Sofia
  - Clincal Site, Stara Zagora
  - Clinical Site, Varna
- France (5):
  - Clinical Site, Douai
  - Clinical Site, Nantes
  - Clinical Site, Nîmes
  - Clinical Site, Paris
  - Clinical Site, Poitiers
- India (9):
  - Clinical Site, Ahmedabad, Gujarat
  - Clinical Site, Rajkot, Gujarat
  - Clinical Site, Surat, Gujarat
  - Clinical Site, Kolhāpur, Maharahstra
  - Clinical Site, Bārāmati, Maharashtra
  - Clinical Site, Nagpur, Maharashtra
  - Clinical Site, Pune, Maharashtra
  - Clinical Site, Wardha, Maharashtra
  - Clinical Site, Ajmer, Rajasthan
- Lithuania (2):
  - Clinical Site, Kaunas
  - Clinical Site, Ziegzdriai
- Serbia (6):
  - Clinical Site, Belgrade
  - Clinical Site, Gornja Toponica
  - Clinical Site, Kovin
  - Clinical Site, Kragujevac
  - Clinical Site, Niš
  - Clinical Site, Novi Kneževac
- Spain (4):
  - Clinical Site, Barcelona
  - Clinical Site, Madrid
  - Clinical Site, Sabadell
  - Clinical Site, Zamora

IPD SHARING:
Plan to Share IPD: No